CLINICAL TRIAL: NCT05847283
Title: Dydrogesterone Primed Ovarian Stimulation Versus Fixed Gonadotropin Releasing Hormone Antagonist Protocol for Oocyte Accumulation in Low Ovarian Reserve Patients: A Randomized Controlled Trial
Brief Title: DPOS Versus GnRH Antagonist Protocol for Oocyte Accumulation in Low Ovarian Reserve Patients: An RCT
Acronym: DPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tam Anh TP. Ho Chi Minh General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Nhu H Giang, MD., MCE., Tam Anh TP. Ho Chi Minh General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DYDR-C22-0313
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diminished Ovarian Reserve
Keywords: Progestin priming ovarian stimulation; Oocyte accumulation; Diminished ovarian reserve; GnRH antagonist; Oocyte vitrification; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPOS protocol (Active Comparator): Women will receive oral Dydrogesterone 10mg (Duphaston 10mg) t.i.d daily from the first day of ovarian stimulation till the day of final oocyte maturation.
  Interventions: Procedure: Dydrogesterone priming ovarian stiumulation protocol
- GnRH antagonist protocol (Placebo Comparator): Women will receive GnRH antagonist (Ganirelix 0.25mg) once subcutaneously daily from day 5 of ovarian stimulation till the day of final oocyte maturation
  Interventions: Procedure: GnRH antagonist protocol

INTERVENTIONS:
Procedure: Dydrogesterone priming ovarian stiumulation protocol — Patients will be co-administered with oral DYG (Duphaston) 30mg/d and Human Menopausal Gonadotrophin (hMG) 225 IU/day (IU/d) via intramuscular injection from menstrual cycle day 2 - 4 (CD2 - CD4) to the day of final oocyte maturation.
  Other Names: DPOS protocol
  Arms: DPOS protocol
Procedure: GnRH antagonist protocol — In the fixed GnRH antagonist protocol, hMG 225 IU will be administered daily from menstrual cycle day 2 - 4 (CD2 - CD4) and s.c. administration of GnRH antagonist (Ganirelix 0.25 mg) will be initiated daily on the 5th day of stimulation. Treatment with hMG and GnRH antagonist will be continued until the day of final oocyte maturation triggering.
  Other Names: GnRHanta protocol
  Arms: GnRH antagonist protocol

SUMMARY:
One of the barriers in patients with diminished ovarian reserve (DOR) is the significantly reduced number of oocytes resulting in fewer oocytes collected and embryos formed. Many ovarian stimulation strategies have been proposed to improve oocyte or embryo quantity which is oocyte accumulation could be a potential option with a comparable success rate and reasonable cost.

Progestin-primed ovarian stimulation (PPOS) protocol could be suggested as an alternative method of premature Luteinizing hormone (LH) prevention in IVF. It favors segment Assisted Reproductive Technology (ART) cycles such as frozen embryo transfer (FET), oocyte donor, fertility preservation, and oocyte accumulation set. The protocol is more patient-friendly and affordable than the GnRH antagonist regimen regarding LH suppression during ovarian stimulation.

Many PPOS protocols have been proposed in which the three most common agents include Dydrogesterone (DYG), Micronised Progesterone (MIP), and Medroxyprogesterone acetate (MPA). Indeed, DYG seems to have some advantages, including oral administration and safety which has been used in the treatment of threatened abortion. Initial evidence of PPOS protocol suggests that oocyte quantity and quality are comparable with other ovarian stimulation regimens. However, data related to the PPOS protocol has not been well documented, including Dydrogesteron-primed ovarian stimulation (DPOS).

There has not been an RCT with a large sample size and well-designed to provide more substantial evidence. A randomized trial to compare the effectiveness of PPOS and GnRH antagonist protocol in IVF is urgently needed.

DETAILED DESCRIPTION:
Screening for eligibility and randomization

* This trial will be conducted at Tam Anh TP. Ho Chi Minh General hospital, Ho Chi Minh City, Vietnam and Tam Anh General hospital, Ha Noi, Vietnam
* Women who are potentially eligible will be provided information about the trial when IVF treatment is indicated
* Patients will be provided information related to the study together with the informed consent documents. Signed informed consent forms will be obtained by the investigators from all women before the enrolment.
* Women will be randomized (1:1) to either DPOS or GnRH antagonist protocol

Ovarian stimulation

* The patients will be stimulated with the same protocol in all OS cycles after randomization.
* For DPOS arm (Group I): Patients will be co-administered with oral DYG (Duphaston) 30mg/d and Human Menopausal Gonadotrophin (hMG) 225 IU/day (IU/d) via intramuscular injection from menstrual cycle day 2 - 4 (CD2 - CD4) to the day of final oocyte maturation.
* For GnRH antagonist arm (Group II): In the fixed GnRH antagonist protocol, hMG 225 IU will be administered daily from menstrual cycle day 2 - 4 (CD2 - CD4). Daily administration of GnRH antagonist (Ganirelix 0.25 mg) will be initiated on the 5th day of stimulation. Treatment with hMG and GnRH antagonist will be continued daily until the day of final oocyte maturation triggering.

Oocytes retrieval and cryopreservation

* After 36 hours of final maturation injection, all follicles greater than 12mm in diameter will be aspirated.
* Oocyte cryopreservation will be applied to collect at least 7 ± 1 oocytes
* Matured oocytes will be frozen by vitrification (CRYOTEC® Method)

Oocyte thawing and ICSI

* For the last ovarian stimulation cycle, based on the aim to collect at least 7 ± 1 oocytes, the clinician will determine the last ovarian stimulation cycle on the day of final oocyte maturation.
* The frozen oocytes of the previous OS cycle will be thawed; all fresh and frozen oocytes will be fertilized by ICSI.
* The thawing process will follow the CRYOTEC® Method
* ICSI will be used for the fertilization of mature oocytes.

Embryo cryopreservation

* Both the fresh and frozen fertilized oocytes continue to culture in the CXCM medium (Irvine Scientific., USA) to blastocyst.
* Freeze-all strategy is applied in both arms, then the frozen embryo will be transferred in the next cycle.

Endometrium preparation and embryo transfer

* Endometrial preparation with hormonal replacement therapy will be performed. In the following cycle, the endometrium will be prepared using oral estradiol valerate (Valiera®; Laboratories Recalcine) 6 mg/day starting from the second or third day of the menstrual cycle. The endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Cyclogest®; Actavis) 800 mg/day plus dydrogesterone (Duphaston 10mg) at the dose of 10mg twice daily will be started when endometrial thickness reaches 8 mm or more. Elective single blastocyst transfer will be performed.
* Embryos will be thawed on the day of embryo transfer, five or six days after the start of progesterone depending on the day-5 or day-6 embryo, respectively. Embryos will be transferred into the uterine cavity under ultrasound guidance.

Pregnancy test and ultrasound to confirm fetal viability

* A pregnancy test will be performed by measuring the blood beta-hCG level 10 - 11 days after embryo transfer. If the pregnancy test is positive (≥25mIU/mL), the patient is indicated to use exogenous estrogen and progesterone until at least 12 weeks of gestation.
* A pregnancy ultrasound will be performed three weeks after the positive pregnancy test equal to 7 weeks of gestational age.
* The primary endpoint is ongoing pregnancy (11 - 12 weeks of gestation) after the first embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* Woman aged between 18 and 37 years
* AFC ≤ 5 and/or AMH ≤ 1.2 ng/ml
* Agree to perform freeze-all strategy and single frozen blastocyst embryo transfer

Exclusion Criteria:

* Oocyte recipient
* Indication of preimplantation genetic testing
* Known allergic reactions to medications in the Study (progesterone products, GnRH antagonist….)
* Basal FSH above 15mIU/mL.
* Have contraindications of ART treatment (e.g. critical or acute diseases)
* Retrieved sperm
* Repeated Implantation failure ( ≥ 3 failed embryo transfers with good-quality embryos)
* Inability to comply with the study procedures.
* Patients with a history of thyroid cancer who are on hormone replacement therapy or those diagnosed with thyroid diseases at the time of eligibility assessment

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 730 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate after the first embryo transfer | 11 - 12 weeks of gestation
  Ongoing pregnancy is defined as pregnancy with a detectable heart rate at 11 - 12 weeks of gestation after the completion of the first transfer.

SECONDARY OUTCOMES:
Serum LH level | On day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
  LH levels are measured on day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
Serum Estradiol level | On day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
  Estradiol levels are measured on day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
Serum Progesterone level | On day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
  Progesterone levels are measured on day 1, day 5, day 8 of FSH administration, on the trigger day and 12 hours after the trigger injection
Premature LH surge | on the day of trigger, an average of 2 weeks after FSH administration
  Premature LH surge (PLS) is increased serum LH more than twice the baseline or more than 15 mIU/ml. The rate of Premature LH surge is defined as number of PLS appearances per number of ovarian stimulation cycles
Duration of ovarian stimulation | From the day 1 of FSH administration to the day of trigger, an average of 2 weeks after FSH administration
  Number of ovarian stimulation days
Total dose of FSH | From the day 1 of FSH administration to the day of trigger, an average of 2 weeks after FSH administration
  A number of international units of FSH are administrated during an ovarian stimulation cycle
Number of Cumulus-oocyte complex | On the oocyte retrieval day, an average of 2 weeks after FSH administration
  Number of Cumulus-oocyte complexes after oocyte retrieval
Number of MII oocyte | On the oocyte retrieval day, an average of 2 weeks after FSH administration
  Number of MII oocytes after denuding
Number of survival oocyte | On the oocyte retrieval day of the ovarian stimulation cycle for ICSI, an average of 2 weeks after FSH administration
  Number of survival oocytes after thawing
Fertilization rate per oocyte inseminated/injected | On the oocyte retrieval day of the ovarian stimulation cycle for ICSI, an average of 2 weeks after FSH administration
  Fertilization is defined as the appearance of two PN at 17±1 hour per inseminated/injected
Embryo-cleavage rate | Day 3 after ICSI day
  Number of embryos on Day 3 after ICSI day
Blastocyst rate | Day 5 and Day 6 after ICSI day
  Numbers of embryos on Day 5 and Day 6 after ICSI
Number of survival blastocyst | Day 5 and Day 6 after ICSI day
  Number of survival embryos on Day 5 and Day 6 after thawing
Top-quality blastocyst rate | Day 5 and Day 6 after ICSI day
  Numbers of embryos on Day 5 and Day 6 with good quality after ICSI
Positive pregnancy test | 11 days after the first transfer
  A positive pregnancy test is defined as a serum hCG level greater than 25 mIU/mL 11 days after the first transfer
Implantation rate | Within 12 weeks of gestation
  Implantation rate is defined as the number of gestational sacs per number of embryos transferred 3 weeks after the first transfer
Biochemical pregnancy | Within 12 weeks of gestation
  Biochemical pregnancy is defined as a pregnancy diagnosed only by the detection of beta hCG in serum or urine
Miscarriage | Within 12 weeks of gestation
  Complete loss of clinical pregnancy at 12 weeks of gestation
Multiple pregnancy rate | Within 12 weeks of gestation
  Multiple pregnancy rate is explained as two or more gestational sacs or positive heartbeats by transvaginal sonography 5 weeks after embryo placement
Ectopic pregnancy rate | Within 12 weeks of gestation
  Ectopic pregnancy confirmed by sonography or laparoscopy at 12 weeks of gestation
Adverse events | Through study completion of each individual patient, an average of 6 months
  Adverse events regarding medications according to local information products
Drop-out | Through study completion, approximately within 2 years
  Drop-out is defined as any patient discontinuing the Study or the investigator withdrawing them from the Study for any reason.
Quality of life score | On day 1 of FSH administration of the first ovarian stimulation cycle for oocyte vitrification and on the trigger day of the ovarian stimulation cycle for ICSI
  Quality of life is assessed by Vietnamese WHO-BRIFE questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nhu H Giang, MD., MCE, Principal Investigator — Tam Anh TP. Ho Chi Minh General Hospital
Locations (2):
- Vietnam (2):
  - IVFTA, Hanoi, Hanoi
  - Ivfta Hcmc, Ho Chi Minh City, Ho Chi Minh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT05847283/Prot_001.pdf